CLINICAL TRIAL: NCT06150157
Title: A First-in-Human Study of the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-88549968, a T-cell Redirecting Bispecific Antibody for CALR-mutated Myeloproliferative Neoplasms
Brief Title: A Study of JNJ-88549968 for the Treatment of Calreticulin (CALR)-Mutated Myeloproliferative Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 88549968MPN1001; 88549968MPN1001 (Other: Janssen Research & Development, LLC); 2023-505584-36-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Myeloproliferative Disorders; Essential Thrombocythemia; Neoplasms; Myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombocythemia, Essential; Neoplasms; Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dose Escalation (Part 1) and Dose Expansion (Part 2) (Experimental): In dose escalation (Part 1), participants will receive JNJ-88549968. The dose will be escalated sequentially to determine the recommended phase 2 dose (RP2D) and optimal dosing schedule(s) based on safety, pharmacokinetic, pharmacodynamic, and preliminary assessment of efficacy across several dose regimens. In dose expansion (Part 2), participants will receive JNJ-88549968 at the RP2D regimen(s) determined in dose escalation (Part 1).
  Interventions: Drug: JNJ-88549968; Drug: Ruxolitinib

INTERVENTIONS:
Drug: JNJ-88549968 — JNJ-88549968 will be administered.
Drug: Ruxolitinib — For US sites: Ruxolitinib will be administered for participants with MF only.

SUMMARY:
The purpose of this study is to characterize safety and to determine the Recommended Phase 2 Dose (RP2D[s]) and optimal dosing schedule(s) of JNJ-88549968, in part 1 (Dose Escalation); to characterize the safety of JNJ- 88549968 at RP2D(s), in part 2 (Cohort Expansion).

ELIGIBILITY:
Inclusion Criteria:

* Be greater than or equal to (>=) 18 years of age (or the legal age of majority in the jurisdiction in which the study is taking place, whichever the greater) at the time of informed consent
* Positive for a calreticulin (CALR) driver mutation of essential thrombocythemia (ET) or myelofibrosis (MF)
* Participants with ET and MF with risk characteristics as described in the protocol
* Have an Eastern Cooperative Oncology Group (ECOG) performance status grade of less than or equal to (<=) 2

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to the excipients of the study treatment
* Concurrent or recently diagnosed or treated malignancies present at the time of participant screening. Exceptions are squamous and basal cell carcinoma of the skin, carcinoma in situ of the cervix, and any malignancy that is considered cured or has minimal risk of recurrence within 1 year of first dose of study treatment in the opinion of both the investigator and sponsor's medical monitor. Participants cured of another malignant disease with no sign of relapse greater than or equal to (>=) 3 years after treatment ended are allowed to enter the study
* Prior solid organ transplantation
* Either of the following regarding hematopoietic stem cell transplantation:

  1. Prior treatment with allogenic stem cell transplant less than or equal to (<=) 6 months before the first dose of JNJ-88549968 or
  2. Evidence of graft versus host disease (GVHD) that requires immunosuppressant therapy
* History of clinically significant cardiovascular disease within 6 months prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-12-04 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Dose Limiting Toxicity (DLT) | Approximately up to 35 days after first dose of study treatment
  Number of participants with DLT will be reported. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Part 1 and 2: Number of Participants with Adverse Events (AEs) | Up to 2 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Part 1 and 2: Number of Participants with Adverse Events (AEs) by Severity | Up to 2 years
  An adverse event is any untoward medical occurrence in a clinical study participant that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from grade 1 (mild) to grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to adverse event. Cytokine release syndrome (CRS) and associated neurologic toxicity events (immune effector cell-associated neurotoxicity syndrome events [ICANS]) will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines.

SECONDARY OUTCOMES:
Part 1 and 2: Serum Concentration of JNJ-88549968 | Up to 2 years
  Serum samples will be analyzed to determine concentrations of JNJ-88549968.
Part 1 and 2: Number of Participants With Presence of Anti-Drug Antibodies to JNJ-88549968 | Up to 2 years
  Number of participants with presence of anti-drug antibodies to JNJ-88549968 will be reported.
Part 1 and 2: Overall Response Rate | Up to 2 years
  ORR is defined as the percentage of participants who achieve partial response (PR) and complete response (CR) according to modified International Working Group-Myeloproliferative Neoplasm Research and Treatment (IWG-MRT) criteria and modified European Leukemia Net (ELN) consensus report.
Part 1 and 2: Complete Response (CR) Rate | Up to 2 years
  CR rate is defined as the percentage of participants who achieve a best response of CR according to disease as defined in modified IWG-MRT criteria and modified ELN consensus report.
Part 1 and 2: Time to Response (TTR) | Up to 2 years
  TTR is defined for participants who achieved PR or CR as the time from the first dose of study treatment to first response of PR or CR according to modified IWG-MRT criteria and modified ELN consensus report.
Part 1 and 2: Duration of Response (DOR) | Up to 2 years
  DOR is defined for participants who achieved PR or CR as the time between the date of initial documentation of PR or CR to the date of first documented evidence of disease progression, as defined in modified IWG-MRT criteria and modified ELN consensus report, or death, whichever comes first.
Part 2: Change From Baseline in Myeloproliferative Neoplasm (MPN) Symptom Burden | Baseline up to 2 years
  Change from baseline in MPN symptom burden assessed using patient reported outcome (PRO) questionnaire will be reported in this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (29):
- United States (8):
  - City of Hope, Duarte, California
  - Moffit Cancer center, Tampa, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Cancer Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (2):
  - Hopital Saint Louis, Paris
  - CH LYON SUD - Hematology, Pierre-Bénite
- Germany (6):
  - Universitaetsklinikum der RWTH Aachen, Aachen
  - Charite Campus Benjamin Franklin, Berlin
  - Med. Universitatsklinik Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Regensburg, Regensburg
- Israel (4):
  - Carmel Medical Center, Haifa
  - Hadassah University Hospita Ein Kerem, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Policlinico di Milano, Milan
- Spain (2):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Clinico Univ. de Valencia, Valencia
- United Kingdom (3):
  - University College London Hospitals Nhs Foundation Trust, London
  - Guy's and St Thomas' Hospital, London
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency